CLINICAL TRIAL: NCT01424176
Title: A Multicenter, Open-Label, Single-dose, Pharmacokinetic and Safety Study of Dexpramipexole (BIIB050) in Healthy Subjects and Subjects With Renal Impairment
Brief Title: Dexpramipexole Renal PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 223RI101
Record Dates: First submitted 2011-06-23; First posted 2011-08-26 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Renal Insufficiency
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Renal Insufficiency | interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexpramipexole (dose 1) (Experimental): Subjects with mild or moderate renal impairment.
  Interventions: Drug: Dexpramipexole (dose 1)
- Dexpramipexole (dose 2) (Experimental): Subjects with severe renal impairment and end stage renal disease (ESRD).
  Interventions: Drug: Dexpramipexole (dose 2)

INTERVENTIONS:
Drug: Dexpramipexole (dose 1)
  Other Names: BIIB050
  Arms: Dexpramipexole (dose 1)
Drug: Dexpramipexole (dose 2)
  Other Names: BIIB050
  Arms: Dexpramipexole (dose 2)

SUMMARY:
This is a multicenter, open-label, single-dose, PK and safety study in subjects with various stages of renal impairment.

DETAILED DESCRIPTION:
Dexpramipexole (BIIB050, KNS-760704; (6R)-4,5,6,7-tetrahydro-N6-propyl-2,6-benzothiazolediamine dihydrochloride monohydrate) is a synthetic amino-benzothiazole. Data from multiple in vitro and in vivo assays have suggested that dexpramipexole is neuroprotective. It is being investigated for the treatment ALS.

As dexpramipexole is principally eliminated from the body by the kidneys a single oral dose of dexpramipexole will be administered to subjects with various stages of renal impariment comprising the following categories: mild, moderate, severe and ESRD subjects. Healthy volunteers will be matched to each catergory of renal impaired subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/females aged 18 to 75 years inclusive and between 19 and 36 kg/m2 inclusive BMI.
* Subjects with renal impairment must have stable renal disease (i.e., no change in disease status within the 28 days prior to dosing) as determined by the Investigator with laboratory and clinical findings that support the diagnosis of renal impairment.
* Subjects with renal impairment (excluding ESRD subjects), must have 2 separate estimates of creatinine clearance that are within 25% of each other, obtained >5 days apart, but not >6 months apart
* Subjects must have a GFR (estimated GFR; as defined by estimation of creatinine clearance using the MDRD formula) of ≥80 (healthy volunteers), between 50 and 79 (mild renal impairment), between 30 and 49 (moderate renal impairment), or <30 (severe renal impairment), or must require dialysis ≤3 times a week (ESRD).
* Healthy volunteers must be matched to renally impaired subjects for age (± 10 years), gender, and if possible BMI (± 20%).

Exclusion Criteria:

* Healthy volunteers who have received prescription medication within the 14 days prior to dosing (except for birth control).
* Renally impaired subjects who have received prescription medication within the 14 days prior to dosing (except for birth control and medications taken at a stable dose for underlying conditions, as determined by the Investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
AUC after single dose of dexpramipexole | pre dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours after dosing in all subjects, and in addition at 96, 120, and 144 hours after dosing in subjects with severe renal impairment and ESRD.
Cmax after single dose of dexpramipexole | pre dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours after dosing in all subjects, and in addition at 96, 120, and 144 hours after dosing in subjects with severe renal impairment and ESRD.

SECONDARY OUTCOMES:
Mointoring of Clinical Laboratory tests | pre-144 hours post dose
ECG Monitoring | pre-144 hrs post dose
Vital Sign monitoring | pre-144 hrs post dose
AE monitoring | pre-144 hrs post dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Orlando, Florida
  - Research Site, Brooklyn Center, Minnesota